CLINICAL TRIAL: NCT05284604
Title: A Pilot Study of Mesenchymal Stem Cells as Novel Therapy for Age-Related Frailty in Veterans
Brief Title: Mesenchymal Stem Cells for Age-Related Frailty
Acronym: MESCAFY
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E4096-P
Record Dates: First submitted 2022-03-08; First posted 2022-03-17 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Frailty
Keywords: Frailty; Aging; Mesenchymal Stem Cells; Physical Function; Cognitive Function; Sarcopenia; Osteoporosis
MeSH Terms: conditions — Frailty; Sarcopenia; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of three groups in parallel for the duration of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All investigators, study assessors, and participants will not be aware of the group assessments (double-blinded randomized controlled trial)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1 (Experimental): Peripheral IV Infusion of 100 million MSCs at baseline and repeated at three months
  Interventions: Drug: Mesenchymal Stem Cells (MSCs)
- Group 2 (Experimental): Peripheral IV Infusion of 100 million MSCs at baseline and peripheral IV infusion of placebo at three months
  Interventions: Drug: Mesenchymal Stem Cells (MSCs)
- Group 3 (Placebo Comparator): Peripheral IV infusion of placebo at baseline and repeated at three months
  Interventions: Drug: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Drug: Mesenchymal Stem Cells (MSCs) — The MSCs are recovered from bone marrows of healthy donors. Each donor is carefully screened for pathogens to assure the product is safe. The MSCs are strictly compliant with FDA standards under Current Good Manufacturing Practice (cGMP) regulations.

SUMMARY:
Frailty is a health state related to the aging process in which multiple body systems gradually lose their built-in reserves. It is a medical condition of reduced function in older adults which is associated with increased risks of adverse outcomes such as falls, disability, admission to hospital, or need for long-term care. Currently, there is no specific medical treatment of frailty. Mesenchymal stem cells (MSCs) are undifferentiated cells that self-replicated, and some may change into a particular cell type. These cells go to areas of injury due to signals released by injured cells. Upon reaching, the target tissue, MSCs repair injury by releasing growth factors and immune modulators to assist in the body's repair process. This initial study will assess the practicability of using MSCs for age-related frailty and provide information for planning a future full study of MSCs for maximizing Veteran's functional independence.

DETAILED DESCRIPTION:
Frailty is an aging-related syndrome of impaired physiologic reserve and function across multiple organs, leading to increased vulnerability for adverse health outcomes. Frailty is associated with an increased risk for falls, disability, hospitalization, and mortality. Given the rapid growth in the aging population, the prevalence of frailty will continue to increase. In fact, Veterans receiving care at Veterans Health Administration are a high risk population for onset of frailty due to being predominantly older associated with a larger proportion of minorities, lower socioeconomic and educational status, higher prevalence of comorbidities, and higher rates of unemployment. Frailty now affects at least 3 of every 10 U.S. Veterans aged 65 years and older and is strongly associated with mortality. It is increasingly being recognized that frailty may be an appropriate target for intervention to reduce disability and dependence in older adults. However, there are no specific medical or biologic treatments that ameliorate or reverse frailty. Conversely, stem cell depletion is a key mechanism for age-related frailty. There is a strong link between frailty, inflammation, and the impaired ability to repair tissue injury due to decreases in endogenous stem cell production. Accordingly, a cell-based, regenerative treatment strategy i.e., allogenic bone-marrow derived mesenchymal stem cell (MSC) therapy may represent a novel therapy for aging frailty. MSCs migrate into the site of injury and home to the affected tissue, where they act to reduce inflammation and promote cellular repair. The advantages of MSCs as a therapeutic strategy for age-related frailty include availability, ease of isolation and expansion, multilineage differentiation and immunosuppression, free from ethical issues, and limited replicative lifespan. In this 6-month pilot study, the investigators will assess 1) the feasibility of MSC therapy in age-related frailty as it relates to functional improvement and 2) develop/refine MSC therapy as a new intervention in older Veterans with frailty, and thus provide preliminary participant response to inform a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 - 85 years and living in the community
* Modified Physical Performance Test score of 18 to 31
* Clinical Frailty Scale score of 5 or 6
* 6-minute walk distance of >200m and <400m
* Willing to provide informed consent

Exclusion Criteria:

* Failure to provide informed consent
* Major cardiopulmonary disease (e.g., recent MI, unstable angina, stroke) or unstable disease (e.g. NYHA Class II or IV congestive heart failure, severe pulmonary disease requiring steroid pills or the use of supplemental oxygen
* Severe neuromuscular disease (e.g., multiple sclerosis, Parkinson's disease, Amyotrophic lateral sclerosis)
* Renal impairment as defined by an estimated glomerular filtration rate (eGFR or less than 30 ml/min/1.73 m2)
* Other significant co-morbid disease (e.g., severe psychiatric disorder [e.g. bipolar, schizophrenia], excess alcohol use (>14 drinks per week)
* Uncontrolled hypertension (BP>160/90 mm Hg)
* Significant cognitive impairment, defined as a known diagnosis of dementia or positive screening test for dementia using the Mini-Mental State Exam (i.e., MMSE score <24)
* Poorly controlled diabetes (HbA1c >8.5%)
* History of malignancy during the past 5 years (except non-melanoma skin cancers)
* Have autoimmune disease (e.g., Rheumatoid arthritis, systemic lupus erythematosus)
* Be using chronic immunosuppressant therapy such as high-dose corticosteroids or TNF-alpha antagonists (prednisone use at doses of < 5 mg daily is allowed)
* Test positive for hepatitis B virus - If the subject tests positive for anti-hepatitis B core antigen (HBc) or anti-HBs, they must be currently receiving treatment for Hepatitis B prior to infusion and remain on treatment throughout the study
* Test positive for Hepatitis C virus, HIV1/2, or syphilis
* Have any clinically important screening laboratory values, including hemoglobin <10.0 g/dL, WBC <2.500/ul or platelet count<100,000/ul, AST or ALT > 3 times the upper limit of normal, INR>1.3 not due to reversible cause (e.g., warfarin)
* Treatment with another investigational drug or other intervention within three months
* A history or current evidence of any condition, laboratory abnormality, or other circumstance that might confound the interpretation of the results

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence | Through study completion at 6 months
  Percent of study visits attended

SECONDARY OUTCOMES:
Recruitment | Through study completion at 6 months
  Number of participants recruited
Modified Physical Performance Test | Change from baseline to 6 months
  Includes seven standardized tests (walking 15.2 m, putting and removing a coat, picking up a penny, standing up from a chair, lifting a book, climbing one flight of stairs, and progressive romberg test) plus two additional tasks (going up and down four flights of stairs and making a 360-degree turn). Perfect score is 36
6-Minute Walk Test | Change from baseline to 6 months
  A performance based measure of functional exercise capacity.

OTHER OUTCOMES:
4-minute walk gait speed | Change from baseline to 6 months
  Time needed to walk 4 meters at the usual pace will be measured
Activities of daily living (ADL) and instrumental ADL | Change from baseline to 6 months
  Assessed using the physical function subscale of the Functional Status Questionnaire
High-Sensitivity C-reactive protein | Change from baseline to 6 months
  Marker of chronic inflammation - measured by immunoturbidimetric assay
Knee extensor strength | Change from baseline to 6 months
  as evaluated using a Biodex System 3 dynamometer
Soluble tumor necrosis factor receptor 1 (sTNF) | Change from baseline to 6 months
  Measured in serum using enzyme-linked immunoabsorbent assay
Interleukin-6 | Change from baseline to 6 months
  Measured in serum using enzyme-linked immunoabsorbent assay
Bone mineral density of the lumbar spine and hip | Change from baseline to 6 months
  Measured using dual-energy x-ray absorptiometry
Lean body mass | Change from baseline to 6 months
  Measured by dual-energy x-ray absorptiometry
Visceral fat mass | Change from baseline to 6 months
  Measured by dual-energy x-ray absorptiometry (DXA)
Bone microarchitecture | Change from baseline to 6 months
  Measured by High-resolution peripheral computed tomography (HR-pQCT) at wrist and distal radius
Bone strength | Change from baseline to 6 months
  Measured using micro-finite element analyses of HR-pQCT
Trabecular bone score | Change from baseline to 6 months
  A textual parameter that provides an index of trabecular microarchitecture
Cognition | Change from baseline to 6 months
  Using the Composite Age-Adjusted Scale Score from the National Institute of Health Toolbox Cognition Battery.
Quality of Life | Change from baseline to 6 months
  Using the Physical a nd Mental component subscale of the Medical Outcomes Study SF-36
Body fat | Change from baseline to 6 months
  Measured using dual-energy x-ray absorptiometry
Grip strength | Change from baseline to 6 months
  Evaluated with a Jamar Handheld dynamometer
Adverse Events | Through study completion at 6 months
  Number of non-serious and serious adverse events
Short Physical Performance Battery | Change from baseline to 6 months
  Objective assessment tool for evaluating lower extremity function
Lipoprotein levels | Change from baseline to 6 months
  Measured using automated enzymatic/colorimetric assays

CONTACTS AND LOCATIONS:
Overall Officials: Dennis T Villareal, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
MEDVAMC will not provide unrestricted, open public access to large scale health related datasets because of re-identification concerns and the obligation to protect Veterans' private information. However, controlled public access will be provided to the greatest extent possible under specific DUAs or other written agreements, and open access will be provided to the final datasets underlying peer-reviewed publications (aggregated data that can be released with privacy and confidentiality risks).